CLINICAL TRIAL: NCT02047318
Title: A Multicentre Extension Study to Evaluate the Long-Term Safety and Durability of the Therapeutic Effect of LUM001 Also Known as Maralixibat (MRX), an Apical Sodium-Dependent Bile Acid Transporter Inhibitor (ASBTi), in the Treatment of Cholestatic Liver Disease in Pediatric Subjects With Alagille Syndrome
Brief Title: An Extension Study to Evaluate the Long-Term Safety and Durability of Effect of LUM001 in the Treatment of Cholestatic Liver Disease in Subjects With Alagille Syndrome (ALGS)
Acronym: IMAGINE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUM001-303; 2013-003832-54 (EudraCT Number)
Record Dates: First submitted 2014-01-23; First posted 2014-01-28 (Estimated); Results first posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Alagille Syndrome
MeSH Terms: conditions — Alagille Syndrome | interventions — maralixibat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LUM001 (Maralixibat) (Experimental): LUM001 also known as Maralixibat (MRX) administered orally up to twice each day
  Interventions: Drug: LUM001 (Maralixibat)

INTERVENTIONS:
Drug: LUM001 (Maralixibat) — Dosing of LUM001 also known as Maralixibat (MRX) with the objective of achieving optimal control of pruritus at a dose level that is tolerated by the participant and up to a maximum daily dose of 560 micrograms per kilogram (mcg/kg).

SUMMARY:
The purpose of this extension study is to determine the long-term safety and tolerability of an investigational treatment (LUM001 also known as Maralixibat) in children with ALGS who have completed participation in a core LUM001 treatment protocol. Efficacy will be assessed by evaluating the effect of LUM001 on pruritus, biochemical markers of pruritus, as well as biochemical markers of cholestasis and liver disease.

ELIGIBILITY:
Participation for an individual patient is expected to be approximately 72 weeks.

Patients who complete 72 weeks of treatment may be eligible to receive treatment for up to 52 weeks during the follow-up treatment period and patients who completed the 124 weeks of treatment may be eligible to enter the additional long-term follow-up period.

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2013-12-20 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2020-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Mirum
Locations (3):
- United Kingdom (3):
  - Birmingham Children's Hospital, Birmingham, West Midlands
  - Leeds Teaching Hospital NHS Trust, Leeds, West Yorkshire
  - Kings College Hospital, London

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants within the study were enrolled from the lead-in Study LUM001-302, where they received various doses of maralixibat (LUM001, MRX) or placebo. Within this study, after a short dose escalation period, participants received MRX 280 ug/kg/day, which consisted of the majority of their exposure within the study. As such, summaries are presented as a single arm, MRX.
Period: Core Study Period
Arm/Group | LUM001 (Maralixibat)
Started | 19
Received MRX 14 ug/kg/Day (Only participants who received PBO in the previous study, LUM001-302, went through dose escalation.) | 6
Received MRX 35 ug/kg/Day (Only participants who received PBO in the previous study, LUM001-302, went through dose escalation.) | 6
Received MRX 70 ug/kg/Day (Only participants who received PBO in the previous study, LUM001-302, went through dose escalation.) | 6
Received MRX 140 ug/kg/Day (Only participants who received PBO in the previous study, LUM001-302, went through dose escalation. Additionally, participants who were randomized to receive 140 ug/kg/day in LUM001-302 were kept at their previous dose when entering this study.) | 11
Received MRX 280 ug/kg/Day (All participants reached the 280 ug/kg/day dose, either through dose escalated or by continuing their previous dose from LUM001-302.) | 19
Completed | 7
Not Completed | 12
Not completed — Did not consent to 52-week follow- up | 8
Not completed — Adverse Event | 1
Not completed — Withdrawal by caregiver | 3
Period: 52-week Follow-up Treatment Period
Arm/Group | LUM001 (Maralixibat)
Started | 6
Completed | 6
Not Completed | 0
Period: Long-term Follow-up Treatment Period
Arm/Group | LUM001 (Maralixibat)
Started | 7
Received MRX 280 ug/kg/Day | 7
Received 420 ug/kg/Day (Participants who received 420ug/kg/day, received 280ug/kg dose in the morning and 140ug/kg in the afternoon during the long term extension period.) | 5
Received 560 ug/kg/Day (Participants who received 560ug/kg/day, received 280ug/kg dose in the morning and 280ug/kg in the afternoon during the long term extension period.) | 5
Completed | 6
Not Completed | 1
Not completed — consent withdrawn by subject | 1

BASELINE CHARACTERISTICS:
Population: After a short dose escalation period, participants received MRX 280 ug/kg/day, which consisted of most of their exposure within the study. As such, summaries are presented as a single arm, MRX.
Groups:
- Core Study Period: In the lead-in Study LUM001-302, participants were randomized to receive either placebo or active drug (MRX). The last observation obtained before first dose of MRX (either for participants who received MRX in Study LUM001-302 or in Study LUM001-303 for participants who received placebo in Study LUM001-302) was used as the MRX baseline observation for all calculations of change from MRX baseline. For participants who were assigned MRX in Study LUM001-302, results at each post-baseline analysis visit included up to 13 more weeks of treatment than participants who were assigned placebo in Study LUM001-302. The core study period of Study LUM001-303 was from Day 1 to Week 72. It encompassed: - a 4-week double-blind dose-escalation period - an 8-week dose-optimization period - a 60-week stable dosing period. Participants could consent to continued long-term follow-up. The furthest analysis timepoint reached by any participant was Week 336. All participants received MRX.
Arm/Group | Core Study Period
Number analyzed (Participants) | 19
Age, Customized [Number; unit: Subjects]
  <2 years | 3
  2 to 4 years | 6
  5 to 8 years | 5
  9 to 12 years | 2
  13 to 18 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From MRX Baseline to Week 48 in Fasting sBA Levels
Description: The primary endpoint of this study was the mean change from MRX baseline to Week 48 in fasting sBA level.
Time Frame: MRX baseline to Week 48
Population: Data collected from 19 participants at MRX baseline. Data collected at Week 48 from 17 of the 19 participants who contributed values at MRX baseline.
  Since all participants escalated to MRX 280 ug/kg/day by Week 48, the summary is presented as a single arm.
Measure: Mean (Standard Deviation); unit: μmol/L
Groups:
- Core Study Period: MRX Baseline Values: These are the MRX baseline values for participants. The last observation obtained before the first dose of MRX (whether before receiving MRX in Study LUM001-302 for participants who received MRX in Study LUM001-302, or in Study LUM001-303 for participants who received placebo in Study LUM001-302) was used as the MRX baseline observation for all calculations of change from MRX baseline. For participants who were assigned MRX in Study LUM001-302, results at each post-baseline analysis visit included up to 13 more weeks of treatment than participants who were assigned placebo in Study LUM001-302.
- Core Study Period: Week 48 Values: These are the Week 48 values for participants. These participants are also represented in the Core study period: MRX baseline values group; the analyses look at the change from MRX baseline to Week 48 in the same participants.
Arm/Group | Core Study Period: MRX Baseline Values | Core Study Period: Week 48 Values
Number analyzed (Participants) | 19 | 17
μmol/L | 261.96 (206.839) | 128.32 (101.742)
Statistical Analysis 1: Comparison: Core Study Period: MRX Baseline Values vs Core Study Period: Week 48 Values; This analysis investigated whether a statistically significant change in sBA levels was observed when comparing MRX baseline to Week 48. The analysis was based on the safety population; Test type: Equivalence — The null hypothesis that the mean change was equal to zero was tested using the Student's t-test to determine if the mean change in sBA levels between MRX baseline and Week 48 was statistically significant; p = 0.0012, Student's t-test — Data for this analysis were obtained from 19 participants at MRX baseline; 17 of those participants contributed Week 48 data; Mean Difference (Net) = -94.4, 95% CI 2-sided [-145.26 to -43.55], Standard Deviation 98.915

2. Secondary Outcome: Change From MRX Baseline Over Time in Fasting sBA Levels
Description: This secondary efficacy endpoint is the mean change from MRX baseline over time in fasting sBA levels. Results reported here are the long-term results.
Time Frame: MRX baseline to End of Treatment (maximum exposure was 336 weeks)
Population: Data collected from 19 participants at MRX baseline. Data collected at Week 252 from all 6 participants who contributed values at MRX baseline. Week 252 was chosen as this was the latest timepoint with more than 5 participants reporting data and was considered representative of values near the end of treatment. Since all participants escalated to MRX 280 ug/kg/day, the summary is presented as a single arm.
Measure: Mean (Standard Deviation); unit: μmol/L
Groups:
- Core Study Period: MRX Baseline Value: These are the MRX baseline values for participants. The last observation obtained before the first dose of MRX (whether before receiving MRX in Study LUM001-302 for participants who received MRX in Study LUM001-302, or in Study LUM001-303 for participants who received placebo in Study LUM001-302) was used as the MRX baseline observation for all calculations of change from MRX baseline. For participants who were assigned MRX in Study LUM001-302, results at each post-baseline analysis visit included up to 13 more weeks of treatment than participants who were assigned placebo in Study LUM001-302.
- Week 252 Values: Week 252 values for participants continuing in the study. These participants are also represented in the Core study period: MRX baseline values group; the analyses look at the change from MRX baseline to Week 252 in the same participants.
Arm/Group | Core Study Period: MRX Baseline Value | Week 252 Values
Number analyzed (Participants) | 19 | 6
μmol/L | 261.96 (206.839) | 118.32 (76.140)
Statistical Analysis 1: Comparison: Core Study Period: MRX Baseline Value vs Week 252 Values; This analysis investigated whether a statistically significant change in sBA levels was observed over time (with Week 252 chosen as the end point, as the last analysis visit with at least 6 participants). The analysis was based on the safety population; Test type: Equivalence — The null hypothesis that the mean change was equal to zero was tested using the Student's t-test to determine if the mean change in sBA levels from baseline over time (to Week 252) was statistically significant; p = 0.032, Student's t-test — Data for this analysis were obtained from 19 participants at MRX baseline; 6 of those participants contributed Week 252 data; Mean Difference (Net) = -141.94, 95% CI 2-sided [-265.77 to -18.12], Standard Deviation 117.992

3. Secondary Outcome: Change From MRX Baseline to Week 48 in Pruritus
Description: This secondary efficacy endpoint is the change from MRX baseline to Week 48 in pruritus as measured by ItchRO(Obs) weekly average morning severity score. ItchRO scores range from 0 to 4; the higher score indicates increasing itch severity (0 = none; 4 = very severe).
Time Frame: MRX baseline to Week 48
Population: Values were collected from 19 participants at MRX baseline. Data collected at Week 48 from 17 of the 19 participants who contributed values at MRX baseline.
  Since all participants escalated to MRX 280 ug/kg/day by Week 48, the summary is presented as a single arm.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Core Study Period: MRX Baseline Value | Core Study Period: Week 48 Values
Number analyzed (Participants) | 19 | 17
scores on a scale | 2.435 (0.7952) | 1.307 (0.6995)
Statistical Analysis 1: Comparison: Core Study Period: MRX Baseline Value vs Core Study Period: Week 48 Values; This analysis investigated whether a statistically significant change in ItchRO(Obs) scores was observed when comparing MRX baseline to Week 48. The analysis was based on the safety population; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, Student's t-test — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -1.095, 95% CI 2-sided [-1.464 to -0.726], Standard Deviation 0.7173

4. Secondary Outcome: Change From MRX Baseline Over Time in Pruritus
Description: This secondary efficacy endpoint is the change from MRX baseline over time in pruritus as measured by ItchRO(Obs) weekly average morning severity score. ItchRO scores range from 0 to 4; the higher score indicates increasing itch severity (0 = none; 4 = very severe). Results reported here are the long-term results.
Time Frame: MRX baseline to End of Treatment (maximum exposure was 336 weeks)
Population: Data collected from 19 participants at MRX baseline Data collected at Week 278 from all 6 participants who contributed values at MRX baseline. Week 278 was chosen as this was the latest timepoint with more than 5 participants reporting data and was considered representative of values near the end of treatment. Since all participants escalated to MRX 280 ug/kg/day, the summary is presented as a single arm.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Week 278 Values: Week 278 values for participants continuing in the study.
Arm/Group | Core Study Period: MRX Baseline Value | Week 278 Values
Number analyzed (Participants) | 19 | 6
scores on a scale | 2.435 (0.7952) | 0.952 (0.4302)
Statistical Analysis 1: Comparison: Core Study Period: MRX Baseline Value vs Week 278 Values; This analysis investigated whether a statistically significant change in ItchRO(Obs) scores was observed over time (with Week 158 chosen as the end point, as the last analysis visit with at least 6 participants). The analysis was based on the safety population; Test type: Equivalence — The null hypothesis that the mean change was equal to zero was tested using the Student's t-test to determine if the mean change in ItchRO(Obs) scores from baseline over time (to Week 158) was statistically significant; p = 0.0307, Student's t-test — Data for this analysis were obtained from 19 participants at MRX baseline; 6 of those participants contributed Week 158 data; Mean Difference (Net) = -0.958, 95% CI 2-sided [-1.784 to -0.132], Standard Deviation 0.7868

5. Secondary Outcome: Change From MRX Baseline to Week 48 in Clinician Xanthoma Severity Score
Description: This secondary efficacy endpoint is the mean change from MRX baseline to Week 48 in clinician xanthoma severity scores. It is based on a 0-4 scale to rate the number of lesions present and the degree to which the participant's lesions interfere or limit his or her activities. Clinician xanthoma severity scores range from 0 to 4, with a xanthoma score of zero representing no evidence of xanthomatosis and a score of 4 representing xanthoma so severe that it is disabling. Clinician xanthoma severity scores were not assessed in Study LUM001-302 so mean clinician xanthoma severity score at MRX baseline was calculated from the 5 participants who were assigned to placebo in Study LUM001-302, and analysis of change from MRX baseline is not presented.
Time Frame: MRX baseline to Week 48
Population: Mean MRX baseline scores were calculated from the 5 participants assigned placebo in LUM001-302 who had a baseline value in study LUM001-303. Those assigned to MRX within study LUM001-302 did not have this data collected at baseline.
  Mean MRX Week 48 scores were calculated from 17 participants. Since all participants escalated to MRX 280 ug/kg/day by Week 48, the summary is presented as a single arm.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Core Study Period: MRX Baseline Values | Core Study Period: Week 48 Values
Number analyzed (Participants) | 5 | 17
scores on a scale | 0.4 (0.55) | 0.2 (0.73)

6. Secondary Outcome: Change From MRX Baseline Over Time in Clinician Xanthoma Severity Score
Description: This secondary efficacy endpoint is the mean change from MRX baseline over time (with Week 252 chosen as the end point, as the last analysis visit with at least 6 participants) in clinician xanthoma severity scores. It is based on a 0-4 scale to rate the number of lesions present and the degree to which the lesions interfere or limit activities. Clinician xanthoma severity scores range from 0 to 4, with a score of zero representing no evidence of xanthomatosis and a score of 4 representing xanthoma so severe that it is disabling. Clinician xanthoma severity scores were not assessed in Study LUM001-302 so mean clinician xanthoma severity score at MRX baseline was calculated from the 5 participants assigned to placebo in Study LUM001-302, and analysis of change from MRX baseline is not presented. Results reported here are the long-term results.
Time Frame: MRX baseline to End of Treatment (maximum exposure was 336 weeks)
Population: Mean MRX baseline scores were calculated from the 5 participants assigned placebo in LUM001-302.Mean Week 252 scores were calculated from 6 participants. Week 252 was chosen as this was the latest timepoint with more than 5 participants reporting data and was considered representative of values near the end of treatment. Since all participants escalated to MRX 280 ug/kg/day, the summary is presented as a single arm.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Core Study Period: MRX Baseline Value | Week 252 Values
Number analyzed (Participants) | 5 | 6
scores on a scale | 0.4 (0.55) | 0.2 (0.41)

7. Secondary Outcome: Secondary: Change From MRX Baseline to Week 48 in Alkaline Phosphatase
Description: This secondary efficacy endpoint is the mean change from MRX baseline to Week 48 in ALP.
Time Frame: MRX baseline to Week 48
Population: Data collected from 19 participants at MRX baseline. [Data collected at Week 48 from 17 of the 19 participants who contributed values at MRX baseline. Since all participants escalated to MRX 280 ug/kg/day by Week 48, the summary is presented as a single arm.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Core Study Period: MRX Baseline Value | Core Study Period: Week 48 Values
Number analyzed (Participants) | 19 | 17
U/L | 601.5 (232.54) | 596.2 (185.20)
Statistical Analysis 1: Comparison: Core Study Period: MRX Baseline Value vs Core Study Period: Week 48 Values; This analysis investigated whether a statistically significant change in ALP levels was observed when comparing MRX baseline to Week 48. The analysis was based on the safety population; Test type: Equivalence — The null hypothesis that the mean change was equal to zero was tested using the Student's t-test to determine if the mean change in ALP levels between MRX baseline and Week 48 was statistically significant; p = 0.8863, Student's t-test — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 7.4, 95% CI 2-sided [-100.7 to 115.6], Standard Deviation 210.32

8. Secondary Outcome: Change From MRX Baseline Over Time in Alkaline Phosphatase
Description: This secondary efficacy endpoint is the mean change from MRX baseline over time in ALP. Results reported here are the long-term results.
Time Frame: MRX baseline to end of treatment (maximum exposure was 336 weeks)
Population: Data collected from 19 participants at MRX baseline. Data collected at Week 252 from 6 participants who contributed values at MRX baseline. Week 252 was chosen as this was the latest timepoint with more than 5 participants reporting data and was considered representative of values near the end of treatment. Since all participants escalated to MRX 280 ug/kg/day, the summary is presented as a single arm.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Core Study Period: MRX Baseline Value | Week 252 Values
Number analyzed (Participants) | 19 | 6
U/L | 601.5 (232.54) | 430.5 (223.56)
Statistical Analysis 1: Comparison: Core Study Period: MRX Baseline Value vs Week 252 Values; This analysis investigated whether a statistically significant change in ALP levels was observed over time (with Week 252 chosen as the end point as the last analysis visit with at least 6 participants). The analysis was based on the safety population; Test type: Equivalence — The null hypothesis that the mean change was equal to zero was tested using the Student's t-test to determine if the mean change in ALP levels from baseline over time (to Week 252) was statistically significant; p = 0.22, Student's t-test — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -184.3, 95% CI 2-sided [-522.5 to 153.8], Standard Deviation 322.22

9. Secondary Outcome: Change From MRX Baseline to Week 48 in Alanine Aminotransferase
Description: This secondary efficacy endpoint is the mean change from MRX baseline to Week 48 in ALT.
Time Frame: MRX baseline to Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Core Study Period: MRX Baseline Value | Core Study Period: Week 48 Values
Number analyzed (Participants) | 19 | 17
U/L | 130.7 (59.12) | 174.5 (97.28)
Statistical Analysis 1: Comparison: Core Study Period: MRX Baseline Value vs Core Study Period: Week 48 Values; This analysis investigated whether a statistically significant change in ALT levels was observed when comparing MRX baseline to Week 48. The analysis was based on the safety population; Test type: Equivalence — The null hypothesis that the mean change was equal to zero was tested using the Student's t-test to determine if the mean change in ALT levels between MRX baseline and Week 48 was statistically significant; p = 0.0307, Student's t-test — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 51.6, 95% CI 2-sided [5.4 to 97.7], Standard Deviation 89.77

10. Secondary Outcome: Change From MRX Baseline Over Time in Alanine Aminotransferase
Description: This secondary efficacy endpoint is the mean change from MRX baseline over time in ALT levels. Results reported here are the long-term results.
Time Frame: MRX baseline to End of Treatment (maximum exposure was 336 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Core Study Period: MRX Baseline Value | Week 252 Values
Number analyzed (Participants) | 19 | 6
U/L | 130.7 (59.12) | 175.3 (101.17)
Statistical Analysis 1: Comparison: Core Study Period: MRX Baseline Value vs Week 252 Values; This analysis investigated whether a statistically significant change in ALT levels was observed over time (with Week 252 chosen as the end point, as the last analysis visit with at least 6 participants). The analysis was based on the safety population; Test type: Equivalence — The null hypothesis that the mean change was equal to zero was tested using the Student's t-test to determine if the mean change in ALT levels from baseline over time (to Week 252) was statistically significant; p = 0.4934, Student's t-test — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 42.3, 95% CI 2-sided [-105 to 189.7], Standard Deviation 140.41

11. Secondary Outcome: Change From MRX Baseline to Week 48 in Aspartate Aminotransferase
Description: This secondary efficacy endpoint is the mean change from MRX baseline to Week 48 in AST levels.
Time Frame: MRX baseline to Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Core Study Period: MRX Baseline Values | Core Study Period: Week 48 Values
Number analyzed (Participants) | 19 | 17
U/L | 127.6 (60.03) | 142.4 (78.94)
Statistical Analysis 1: Comparison: Core Study Period: MRX Baseline Values vs Core Study Period: Week 48 Values; This analysis investigated whether a statistically significant change in AST levels was observed when comparing MRX baseline to Week 48. The analysis was based on the safety population; Test type: Equivalence — The null hypothesis that the mean change was equal to zero was tested using the Student's t-test to determine if the mean change in AST levels between MRX baseline and Week 48 was statistically significant; p = 0.1571, Student's t-test — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 21.2, 95% CI 2-sided [-9.1 to 51.6], Standard Deviation 58.98

12. Secondary Outcome: Change From MRX Baseline Over Time in Aspartate Aminotransferase
Description: This secondary efficacy endpoint is the mean change from MRX baseline over time in AST levels. Results reported here are the long-term results.
Time Frame: MRX baseline to End of treatment (maximum exposure was 336 weeks)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Core Study Period: MRX Baseline Value | Week 252 Values
Number analyzed (Participants) | 19 | 6
U/L | 127.6 (60.03) | 145.0 (56.50)
Statistical Analysis 1: Comparison: Core Study Period: MRX Baseline Value vs Week 252 Values; This analysis investigated whether a statistically significant change in AST levels was observed over time (with Week 252 chosen as the end point as the last analysis visit with at least 6 participants). The analysis was based on the safety population; Test type: Equivalence — The null hypothesis that the mean change was equal to zero was tested using the Student's t-test to determine if the mean change in AST levels from baseline over time (to Week 252) was statistically significant; p = 0.7815, Student's t-test — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 12.2, 95% CI 2-sided [-94.7 to 119], Standard Deviation 101.84

13. Secondary Outcome: Change From MRX Baseline to Week 48 in Gamma Glutamyltransferase
Description: This secondary efficacy endpoint is the mean change from MRX baseline to Week 48 in GGT.
Time Frame: MRX baseline to Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Core Study Period: MRX Baseline Value | Core Study Period: Week 48 Values
Number analyzed (Participants) | 19 | 17
U/L | 476.9 (376.85) | 440.5 (230.60)
Statistical Analysis 1: Comparison: Core Study Period: MRX Baseline Value vs Core Study Period: Week 48 Values; This analysis investigated whether a statistically significant change in GGT levels was observed when comparing MRX baseline to Week 48. The analysis was based on the safety population; Test type: Equivalence — The null hypothesis that the mean change was equal to zero was tested using the Student's t-test to determine if the mean change in GGT levels between MRX baseline and Week 48 was statistically significant; p = 0.9513, Student's t-test — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -3.9, 95% CI 2-sided [-136.4 to 128.7], Standard Deviation 257.78

14. Secondary Outcome: Change From MRX Baseline Over Time in Gamma Glutamyltransferase
Description: This secondary efficacy endpoint is the mean change from MRX baseline over time in GGT. Results reported here are the long-term results.
Time Frame: MRX baseline to End of Treatment (maximum exposure was 336 weeks)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Core Study Period: MRX Baseline Value | Week 252 Values
Number analyzed (Participants) | 19 | 6
U/L | 476.9 (376.85) | 377.5 (163.10)
Statistical Analysis 1: Comparison: Core Study Period: MRX Baseline Value vs Week 252 Values; This analysis investigated whether a statistically significant change in GGT levels was observed over time (with Week 252 chosen as the end point as the last analysis visit with at least 6 participants). The analysis was based on the safety population; Test type: Equivalence — The null hypothesis that the mean change was equal to zero was tested using the Student's t-test to determine if the mean change in GGT levels from baseline over time (to Week 252) was statistically significant; p = 0.7133, Student's t-test — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -56.7, 95% CI 2-sided [-431.2 to 317.9], Standard Deviation 356.88

15. Secondary Outcome: Change From MRX Baseline to Week 48 in Total and Direct Bilirubin
Description: This secondary efficacy endpoint is the mean change from MRX baseline to Week 48 in total bilirubin and direct bilirubin.
Time Frame: MRX baseline to Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Core Study Period: MRX Baseline Value | Core Study Period: Week 48 Values
Number analyzed (Participants) | 19 | 17
mg/dL
  Total bilirubin | 4.47 (4.837) | 4.25 (5.384)
  Direct bilirubin | 3.80 (3.858) | 3.21 (3.656)
Statistical Analysis 1: Comparison: Core Study Period: MRX Baseline Value vs Core Study Period: Week 48 Values; This analysis investigated whether a statistically significant change in total bilirubin levels was observed when comparing MRX baseline to Week 48. The analysis was based on the safety population; Test type: Equivalence — The null hypothesis that the mean change was equal to zero was tested using the Student's t-test to determine if the mean change in total bilirubin levels between MRX baseline and Week 48 was statistically significant; p = 0.7839, Student's t-test — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.16, 95% CI 2-sided [-1.05 to 1.37], Standard Deviation 2.348
Statistical Analysis 2: Comparison: Core Study Period: MRX Baseline Value vs Core Study Period: Week 48 Values; This analysis investigated whether a statistically significant change in direct bilirubin levels was observed when comparing MRX baseline to Week 48. The analysis was based on the safety population; Test type: Equivalence — The null hypothesis that the mean change was equal to zero was tested using the Student's t-test to determine if the mean change in direct bilirubin levels between MRX baseline and Week 48 was statistically significant; p = 0.5298, Student's t-test — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.66 to 0.35], Standard Deviation 0.982

16. Secondary Outcome: Change From MRX Baseline Over Time in Total and Direct Bilirubin
Description: This secondary efficacy endpoint is the mean change from MRX baseline over time in total bilirubin and direct bilirubin. Results reported here are the long-term results.
Time Frame: MRX baseline to End of Treatment (maximum exposure was 336 weeks)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Core Study Period: MRX Baseline Value | Week 252 Values
Number analyzed (Participants) | 19 | 6
mg/dL
  Total bilirubin | 4.47 (4.837) | 5.05 (6.449)
  Direct bilirubin | 3.80 (3.858) | 3.53 (3.727)
Statistical Analysis 1: Comparison: Core Study Period: MRX Baseline Value vs Week 252 Values; This analysis investigated whether a statistically significant change in total bilirubin levels was observed over time (with Week 252 chosen as the end point as the last analysis visit with at least 6 participants). The analysis was based on the safety population; Test type: Equivalence — The null hypothesis that the mean change was equal to zero was tested using the Student's t-test to determine if the mean change in total bilirubin levels from baseline over time (to Week 252) was statistically significant; p = 0.8218, Student's t-test — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.53, 95% CI 2-sided [-6.31 to 5.24], Standard Deviation 5.505
Statistical Analysis 2: Comparison: Core Study Period: MRX Baseline Value vs Week 252 Values; This analysis investigated whether a statistically significant change in direct bilirubin levels was observed over time (with Week 252 chosen as the end point as the last analysis visit with at least 6 participants). The analysis was based on the safety population; Test type: Equivalence — The null hypothesis that the mean change was equal to zero was tested using the Student's t-test to determine if the mean change in direct bilirubin levels from baseline over time (to Week 252) was statistically significant; p = 0.5549, Student's t-test — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.52, 95% CI 2-sided [-2.62 to 1.58], Standard Deviation 2.001

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are AEs with a start date on or after the first dose of study drug and with a start date prior to the last dose of study drug plus 14 days. Maximum exposure was 336 weeks.
Description: After a short dose escalation period (at dose levels less than 280 ug/kg/day), participants received MRX 280 ug/kg/day. An increase to BID dosing up to 560 mcg/kg/day was permitted during the long-term extension. The majority of exposure within the study was at 280 mcg/kg/day. 4 participants started on 140 mcg/kg/day or higher but had a dose interruption and went through dose escalation from 35 mcg/kg/day up to 280 mcg/kg/day. Thus, the counts for AE are higher than the core period.
Groups:
- 14 Microgram Per Kilogram Per Day (mcg/kg/Day): Participants received LUM001 (also known as Maralixibat or MRX) as an oral solution once daily based on participant's weight. Participants who received placebo in the predecessor study LUM001-302 had their dose escalated starting at 14 microgram per kilogram per day (mcg/kg/day) for one week. This reporting group includes the period of time that participants received 14 mcg/kg/day.
- 35 Microgram Per Kilogram Per Day (mcg/kg/Day): Participants received LUM001 (also known as Maralixibat or MRX) as an oral solution once daily based on participant's weight. Participants who received placebo in the predecessor study LUM001-302 had their dose escalated from 14 to 35 for one week. This reporting group includes the period of time that participants received 35 mcg/kg/day.
- 70 Microgram Per Kilogram Per Day (mcg/kg/Day): Participants received LUM001 (also known as Maralixibat or MRX) as an oral solution once daily based on participant's weight. Participants who received placebo in the predecessor study LUM001-302 had their dose escalated from 35 to 70 microgram per kilogram per day (mcg/kg/day) for one week. This reporting group includes the period of time that participants received 70 mcg/kg/day.
- 140 Microgram Per Kilogram Per Day (mcg/kg/Day): Participants received LUM001 (also known as Maralixibat or MRX) as an oral solution once daily based on participant's weight. Participants who received placebo in the predecessor study LUM001-302 had their dose escalated from 70 to 140 microgram per kilogram per day (mcg/kg/day) for one week. This reporting group includes the period of time that participants received 140 mcg/kg/day.
- 280 Microgram Per Kilogram Per Day (mcg/kg/Day): Participants received LUM001 (also known as Maralixibat or MRX) as an oral solution once daily based on participant's weight. Participants who received placebo in the predecessor study LUM001-302 had their dose escalated from 140 to 280 microgram per kilogram per day (mcg/kg/day) for 8-week dose optimization period and during the stable dosing period for up to 124 weeks. Participants who received MRX in the predecessor study LUM001-302 started on their dose from Week 13 of that study (280 mcg/kg/day or highest tolerated dose). This reporting group includes the period of time that participants received 280 mcg/kg/day.
- 420 Microgram Per Kilogram Per Day (mcg/kg/Day): Participants received LUM001 (also known as Maralixibat or MRX) as an oral solution once daily based on participant's weight. Based on efficacy and safety assessments, participants could receive BID dosing after week 136, starting at 420 microgram per kilogram per day (mcg/kg/day) for 4-week dose escalation period. This reporting group includes the period of time that participants received 420 mcg/kg/day.
- 560 Microgram Per Kilogram Per Day (mcg/kg/Day): Participants received LUM001 (also known as Maralixibat or MRX) as an oral solution once daily based on participant's weight. Participants on BID dosing could have their dose escalated from 480 to 560 microgram per kilogram per day (mcg/kg/day) for the remainder of the study. This reporting group includes the period of time that participants received 560 mcg/kg/day.
- LUM001 MRX Treatment: Participants received LUM001 (also known as Maralixibat or MRX) as an oral solution once daily based on participant's weight. Participants who received placebo in the predecessor study LUM001-302 had their dose escalated from 14, 35, 70, and 140 microgram per kilogram per day (mcg/kg/day) for 4-week dose escalation period. Participants who received maralixibat during study LUM001-302, underwent a mock dose escalation and remained on the dose received at the end of study LUM001-302. During 8-weeks of dose optimization period, drug was adjusted in titrated manner up to 280 mcg/kg/day or highest tolerated dose and dosing was continued to complete the stable dosing and safety monitoring periods for up to 136 weeks of cumulative MRX exposure in this study at this dose level. In the long-term extension, participants could receive BID dosing up to 560 mcg/kg/day for the remainder of the study for up to 336 weeks of cumulative MRX exposure in this study. This reporting group includes all doses of MRX.
Arm/Group | 14 Microgram Per Kilogram Per Day (mcg/kg/Day) | 35 Microgram Per Kilogram Per Day (mcg/kg/Day) | 70 Microgram Per Kilogram Per Day (mcg/kg/Day) | 140 Microgram Per Kilogram Per Day (mcg/kg/Day) | 280 Microgram Per Kilogram Per Day (mcg/kg/Day) | 420 Microgram Per Kilogram Per Day (mcg/kg/Day) | 560 Microgram Per Kilogram Per Day (mcg/kg/Day) | LUM001 MRX Treatment
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/10 | 0/10 | 0/13 | 0/19 | 0/5 | 0/5 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/10 | 1/10 | 0/13 | 6/19 | 0/5 | 1/5 | 6/19
Other Adverse Events (participants affected / at risk) | 3/6 | 6/10 | 3/10 | 10/13 | 18/19 | 3/5 | 5/5 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 14 Microgram Per Kilogram Per Day (mcg/kg/Day) (N=6) | 35 Microgram Per Kilogram Per Day (mcg/kg/Day) (N=10) | 70 Microgram Per Kilogram Per Day (mcg/kg/Day) (N=10) | 140 Microgram Per Kilogram Per Day (mcg/kg/Day) (N=13) | 280 Microgram Per Kilogram Per Day (mcg/kg/Day) (N=19) | 420 Microgram Per Kilogram Per Day (mcg/kg/Day) (N=5) | 560 Microgram Per Kilogram Per Day (mcg/kg/Day) (N=5) | LUM001 MRX Treatment (N=19)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear haemorrhage (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal stoma output decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fibrinous bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Medical device change (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 14 Microgram Per Kilogram Per Day (mcg/kg/Day) (N=6) | 35 Microgram Per Kilogram Per Day (mcg/kg/Day) (N=10) | 70 Microgram Per Kilogram Per Day (mcg/kg/Day) (N=10) | 140 Microgram Per Kilogram Per Day (mcg/kg/Day) (N=13) | 280 Microgram Per Kilogram Per Day (mcg/kg/Day) (N=19) | 420 Microgram Per Kilogram Per Day (mcg/kg/Day) (N=5) | 560 Microgram Per Kilogram Per Day (mcg/kg/Day) (N=5) | LUM001 MRX Treatment (N=19)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 4 (5)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 4 (7) | 10 (26) | 0 (0) | 1 (3) | 11 (40)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (3)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 7 (9) | 0 (0) | 3 (5) | 11 (18)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Malabsorption (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Teething (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 0 (0) | 0 (0) | 5 (7)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 3 (4)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 6 (8) | 0 (0) | 1 (3) | 8 (15)
Biliary tract disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Hepatic lesion (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (3)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (8) | 0 (0) | 1 (1) | 5 (9)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hepatitis infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 7 (18) | 0 (0) | 4 (16) | 8 (36)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (4)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 3 (3) | 4 (8)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 10 (25) | 0 (0) | 0 (0) | 11 (28)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 3 (5)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Drain site complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Limb crushing injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Post procedural fever (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 3 (4)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stoma site erythema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Stoma site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (7) | 0 (0) | 0 (0) | 4 (10)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bilirubin urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood parathyroid hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (2) | 3 (6)
Intracardiac pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urobilinogen urine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin D decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Vitamin E decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 2 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Bone metabolism disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (7) | 0 (0) | 0 (0) | 4 (8)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 0 (0) | 2 (6) | 6 (13)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (3) | 4 (6)
Poor quality sleep (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Taste disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Breath holding (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Enuresis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 8 (16) | 0 (0) | 1 (1) | 10 (21)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 0 (0) | 1 (8) | 3 (16)
Fibrinous bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 6 (6) | 0 (0) | 3 (10) | 7 (18)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Xanthelasma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations of the trial such as small numbers of subjects analyzed or technical problems leading to unreliable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/18/NCT02047318/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/18/NCT02047318/SAP_001.pdf